CLINICAL TRIAL: NCT06171191
Title: Move ARound And Get Active: an Intervention to Optimize 24-hour Movement Behaviours in Preschoolers
Acronym: MARGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Onze Lieve Vrouwziekenhuis Aalst (Other); AZ Jan Palfijn Gent (Other); AZ Alma (Other); Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ONZ-2023-0229
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Parents; Child Behavior; Child Obesity; Physical Inactivity; Sedentary Behavior; Sedentary Time; Sleep; Parenting
Keywords: 24-hour movement behavior; physical activity; sedentary behavior; screen time; sleep; preschooler; parenting
MeSH Terms: conditions — Child Behavior; Pediatric Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Prétest, posttest, follow-up test design. Intervention group receives intervention in between prétest en posttest. Control group receives intervention after follow-up
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group receives intervention between prétest and posttest. Three months after posttest they undergo a follow-up test
  Interventions: Behavioral: Move-ARound And Get Active
- Control group (Other): Waiting group. Control group receives intervention after all test (prétest, posttest and follow-up test)
  Interventions: Behavioral: Move-ARound And Get Active

INTERVENTIONS:
Behavioral: Move-ARound And Get Active — The intervention consists of seven sessions for parents and preschoolers, providing strategies to encourage compliance with the 24-hour movement behavior guidelines for preschoolers of the World Health Organisation.
  Other Names: MARGA

SUMMARY:
In 2019, the World Health Organization established new guidelines for physical activity, sedentary screen time, and sleep for children under 5 years old. Unfortunately, only a few (6%) of preschoolers in Flanders, Belgium, adhere to these guidelines. The aim of this study is to test a health program developed to optimize 24-hour behaviors in preschoolers and encourage more children to follow the guidelines. The program was created using the Intervention Mapping Protocol in collaboration with parents. It consists of seven sessions for parents and preschoolers, providing strategies to encourage compliance with the guidelines. The program's effectiveness will be evaluated through a randomized controlled trial, with the intervention group attending the sessions and the control group receiving the intervention materials at the end of the study.

DETAILED DESCRIPTION:
In 2019, the World Health Organization (WHO) established new guidelines for physical activity, sedentary screen behavior, and sleep in children under 5 years old (WHO, 2019). Unfortunately, only a few (6%) preschoolers in Flanders, Belgium, adhere to these guidelines (De Craemer et al., 2018). The objective of this study is to test a health program developed to optimize 24-hour behaviors in preschoolers and encourage more children to adhere to the guidelines. The program was developed using the Intervention Mapping Protocol, in collaboration with parents (Bartholomew, 2011). The program consists of seven sessions for parents and preschoolers, providing strategies to encourage adherence to the guidelines through parenting skills within the framework of self-determination theory (Di Pasquale et al., 2018). The program will be evaluated through a randomized controlled trial. The intervention group will attend the sessions, while the control group will receive the intervention materials at the end of the study.

Aims:

The primary aim is to analyze the intervention effect on 24-hour movement behaviors:

1. Do more preschoolers comply with the World Health Organization 24-hour movement behavior guidelines?
2. Is there an optimal change in the 24-hour composition of preschoolers (i.e., more physical activity, less screen time, and/or more sufficient sleep relative to each other)?

   The secondary aims are:
3. To analyze the intervention effect on parenting within the self-determination theory: Do parents provide more structure, autonomy support, and positive involvement?
4. Process evaluation of the intervention: Describing fidelity, dose delivered, dose received, reach, and context based on Saunders et al. (2005).

   Patient Recruitment:

   - Group of interest: parents and preschoolers aged 2.5-6 years.

   - Recruitment through care providers

   - Information dissemination through flyers and personal interaction with parents. Active informed consent is required for participation, by signing a informed consent form.

   - Participants are assigned to the intervention or control group based on location. Participants recruited via schools at location X and hospital Y are assigned to the intervention group, while those recruited via schools at location A and hospital B are assigned to the control group.

   - Sample size: max. 200 parent-child dyads

   Data Collection:

   - Measurements are conducted before, after, and 3 months after the end of the sessions in both the intervention and control groups.

   - Measurements include height, weight, waist and hip circumference of the preschoolers, ActiGraph GT3X+ activity monitoring for both child and parent, a diary filled out by parents to support the activity monitor, and a questionnaire on demographic data and parent-related factors (e.g., parenting skills).

   - At the end of each session, parents in the intervention group complete a process evaluation questionnaire based on the framework of Saunders et al. (2005). The control group completes questions regarding the context at the end of the sessions, following the framework of Saunders et al. (2005), e.g., participation in health interventions.

   Intervention Session Content:

   A total of seven sessions are spread over 14 weeks, conducted in groups of 12 parent-child dyads.

   - Session 1: Parent: Information session on 24-hour behavior and parenting skills approached from the self-determination theory.

   Child: Omnisport (athletics, gymnastics, dance, and/or ball sports).

   - Session 2: Parent and child: Week scheduling.
   * Session 3:

   Parent: Discussion group on weekly planning. Child: Omnisport (athletics, gymnastics, dance, and/or ball sports). - Session 4: Parent and child: Movement games. - Session 5: Parent and child: Sleep routine. - Session 6: Parent: Discussion group on sleep routine. Child: Omnisport (athletics, gymnastics, dance, and/or ball sports).

   - Session 7: Parent: Information session on sustainable healthy behavior - persistence and dealing with relapse.

   Child: Omnisport (athletics, gymnastics, dance, and/or ball sports).

   Sessions involving parents are conducted by the leading PhD student, while omnisport for preschoolers is led by master's students from the Faculty of Medicine and Health Sciences at UGent (e.g., Rehabilitation Sciences, Exercise and Sports Sciences, Health Promotion) under her guidance.

   Data Management:

   A Data Management Plan was created using DMPonline.be.

   Data Analyses:

   R software will be used for statistical analyses. Participants need complete data for variables included in the analyses relevant to the specific research aim. Outliers with unrealistic values will be checked, and Little's test will assess whether missing data deviates from Missing Completely At Random (MCAR). Logistic regression models will be applied if necessary to explore relationships between missing values and other recorded variables. To analyze intervention effects, multilevel repeated measures will be used with three levels: time, preschooler, organization (kindergartens/hospitals), adjusted for sex, age, socio-economic status, and session group. Compositional data analyses (CoDA) will be applied to analyze the effect on 24-hour composition. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Preschoolers between 2,5 to 6 years
* One parent per preschooler
* Parent needs to be able to understand, speak, read and write Dutch
* Child needs to be able to understand Dutch
* Child needs to be able to wear accelerometer
* Child needs to by mentally and physically able to comply with the 24-hour movement behavior guidelines
* Parent needs to be mentally able to complete the testing and intervention

Exclusion Criteria:

* Are clear based on the inclusion criteria
* Participants will be excluded form analyses when incomplete data required to answer the research question

Ages: 30 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
24-hour movement behaviour: physical activity, sedentary behaviour and sleep | Results in October 2024
  These behaviours will be assessed with accelerometers (GT3X+), To differentiate sedentary behavior from light physical activity and light physical activity from moderate to vigourous physical activity cut-points of 25 and 420 counts/15 seconds will be used respectively (Evenson et al., 2008; Pate et al., 2006)

SECONDARY OUTCOMES:
Parenting practices | Results in October 2024
  Parenting practices will be assessed within the self-determination theory (Di Pasquale et al., 2018), focusing on providing structure, autonomy support and positive involvement
Process | Results in October 2024
  The process of the intervention will be evaluated based on the framework of Saunders et al. (2005): fidelity, dose delivered, dose received, reach and context will by analysed

CONTACTS AND LOCATIONS:
Overall Officials: Ruth De Bruyne, PhD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - Onze-Lieve-Vrouwenziekenhuis Campus Aalst, Aalst, East-Flanders
  - AZ Alma, Eeklo, East-Flanders
  - AZ Jan Palfijn, Ghent, East-Flanders
  - University Hospital Ghent, Ghent, East-Flanders

IPD SHARING:
Plan to Share IPD: Undecided
This is undecided. There is no further plan available

REFERENCES:
- [Derived] Decraene M, Miatke A, Dumuid D, Cardon G, Verloigne M, De Bruyne R, Verbestel V, De Craemer M. Optimising 24-Hour movement behaviours in preschoolers through parenting practices: an evidence-based intervention study. Int J Behav Nutr Phys Act. 2025 Dec 12. doi: 10.1186/s12966-025-01863-z. Online ahead of print. PMID 41388547